CLINICAL TRIAL: NCT05416502
Title: Prospective Observational Evaluation of the Relationship Between the Rates of Spontaneous Passage of Distal Ureteral Stones and the Diameter of the Most Narrow Part of the Distal Ureter
Brief Title: Prospective Relationship Between the Rates of Spontaneous Passage of Distal Ureteral Stones and the Distal Lumen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hiram's Healthcare and Education Company (Industry)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Other Study IDs: B.30.2.ATA.0.01.00
Record Dates: First submitted 2021-11-16; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Ureter Stone
MeSH Terms: conditions — Ureterolithiasis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Passage Observed: Enrolled patients whose stone and ureter diameters are obtained and their stone passage was successful during the follow-up.
  Interventions: Procedure: Ultrasound
- Passage Not Observed: Enrolled patients whose stone and ureter diameters are obtained and their stone passage was not successful during the follow-up.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Enrolled patients underwent ultrasound scan of kidneys, ureters, and the bladder.

SUMMARY:
Patients (female, male, or queer) with ureteral stones (smaller than 1 cm at the widest diameter of the stone) without pyonephrosis, urinary sepsis, or untraceable pain will be enrolled into the study. Ureteral width at the smallest area of the ureter (in most cases UV junction) will be noted during regular ultrasound scans. The ratio of ureteral width to the stone diameter will be correlated with the spontaneous stone passage.

ELIGIBILITY:
Inclusion Criteria:

Ureteral Stone smaller than 1 cm Volunteer to be enrolled

Exclusion Criteria:

Pyonephrosis Urinary Sepsis Untraceable Pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ureter stones
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Passage | 3 months
  The number of recruited individuals whose ureteral stones are found to be passed by their report and it is confirmed by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared among the following criteria:
  * As allowed to the degree which is allowed by the enrolled patients.
  * As required by the researchers
Supporting Information: Study Protocol, SAP, CSR